CLINICAL TRIAL: NCT03664115
Title: The Effect of Itraconazole on the Clinical Outcomes of Patients With Advanced Non Small Cell Lung Cancer Receiving Platinum Based Chemotherapy
Brief Title: Itraconazole in Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa Waheed Mohamed Mostafa, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00000017585
Record Dates: First submitted 2018-09-01; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Lung Cancer
Keywords: Non small cell lung cancer; itraconazole; mtor inhibition; antiangiogensis; antifungal; anticancer; platinum based chemotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Itraconazole; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Interventional, Randomized, Controlled, Prospective, Open label, Phase II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itraconazole Arm (Experimental): Patients will receive intravenous doses of cisplatin 80 mg/m2 on day 1 plus gemcitabine 1000 mg/m2 on days 1 and 8 every 3 weeks for a maximum of 6 cycles + itraconazole 200 mg oral tablet daily, on a 21-day cycle.
  Alternatively, Carboplatin may be used instead of Cisplatin, Carbplatin AUC 5 DAY 1 only Dose = AUC x (GFR + 25) IV in 250 mL Normal Saline over 30 minutes
  Interventions: Drug: Itraconazole 200 mg; Drug: Chemotherapy
- Control Arm (Active Comparator): Patients will receive intravenous doses of cisplatin 80 mg/m2 on day 1 plus gemcitabine 1000 mg/m2 on days 1 and 8 every 3 weeks for a maximum of 6 cycles.
  Alternatively, Carboplatin may be used instead of Cisplatin, Carbplatin AUC 5 DAY 1 only Dose = AUC x (GFR + 25) IV in 250 mL Normal Saline over 30 minutes
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Itraconazole 200 mg — itraconazole 200 mg oral tablet daily, on a 21-day cycle.
  Arms: Itraconazole Arm
Drug: Chemotherapy — intravenous doses of cisplatin 80 mg/m2 on day 1 plus gemcitabine 1000 mg/m2 on days 1 and 8 every 3 weeks for a maximum of 6 cycles.
  Alternatively, Carboplatin may be used instead of Cisplatin, Carbplatin AUC 5 DAY 1 only Dose = AUC x (GFR + 25) IV in 250 mL Normal Saline over 30 minutes

SUMMARY:
Circulating levels of angiogenic factors have been correlated with aggressive tumor growth, prediction of metastasis and prognosis in a wide range of solid tumors, including non-small cell lung cancer.

Food and Drug Administration (FDA) approved Itraconazole as an anti-angiogenic agent including both Vascular endothelial growth factor (VEGF) and fibroblast growth factor (FGF), and inhibited phosphorylation of the primary angiogenic receptors for these factors in 2007 and also known as an inhibitor of Hedgehog signalling, AKT (protein kinase B)/mechanistic target of rapamycin (mTOR) signaling adding its induction of autophagic cell death function based on cellular and laboratory studies, and allowed its use in phase II trials in prostate, lung and skin cancer.

Itraconazole also interferes directly with mitochondrial Adenosine triphosphate (ATP) production, leading to the activation of the adenosine monophosphate (AMP) -activated protein kinase pathway and subsequent inhibition of mTOR pathway (Head et al., 2015).

Testing Itraconazole on experimental settings was associated also with tumor hypoxia, as proved by induction of tumor-specific expression of Hypoxia-inducible factor 1-alpha (HIF1α), as well as decreased tumor micro-vessel load

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in the United States

The American Cancer Society estimates lung cancer incidence in the United States for 2018 to be about 234,030 and about 154,050 deaths.

In 2012, GLOBOCAN estimated that 1.8 million people were diagnosed with lung cancer, accounting for about 13% of total cancer diagnoses.

Lung cancer death rates declined 45% from 1990 to 2015 among men and 19% from 2002 to 2015 among women. From 2005 to 2014, the rate of new lung cancer cases dropped by 2.5% per year in men and 1.2% per year in women, These differences reflect historical patterns in tobacco use, where women began smoking in large numbers many years later than men, and were slower to quit .

World Health Organization (WHO) divides lung cancer into 2 major classes based on its biology, therapy, and prognosis: non small cell lung cancer (NSCLC) and small cell lung cancer (SCLC).

The NSCLC subtype accounts for 87% of lung cancer cases with its most common types to be adenocarcinomas where it is approximately 40% of lung cancers.

Different factors like age, Performance state, co-morbidities, histology, molecular pathology and last but not least; the patient's preferences should be taken into account along the treatment strategy after a multidisciplinary tumor board discussion, to allow adequate and careful evaluation of the available data to reach the most appropriate management plan and treatment modality for each patient individually (Ung et al., 2016).

Platinum doublets Chemotherapy should be considered in all stage IV and inoperable stage III NSCLC patients with epidermal growth factor receptor (EGFR) and Anaplastic lymphoma kinase (ALK) negative disease, without major comorbidities and Performance state 0-2.

Circulating levels of angiogenic factors have been correlated with aggressive tumor growth, prediction of metastasis and prognosis in a wide range of solid tumors, including non-small cell lung cancer.

Food and Drug Administration (FDA) approved Itraconazole as an anti-angiogenic agent including both Vascular endothelial growth factor (VEGF) and fibroblast growth factor (FGF), and inhibited phosphorylation of the primary angiogenic receptors for these factors in 2007 and also known as an inhibitor of Hedgehog signalling, AKT (protein kinase B)/mechanistic target of rapamycin (mTOR) signaling adding its induction of autophagic cell death function based on cellular and laboratory studies, and allowed its use in phase II trials in prostate, lung and skin cancer.

Itraconazole was proved to be among one of the most potent and selective inhibitors of endothelial cell proliferation.

Itraconazole also interferes directly with mitochondrial Adenosine triphosphate (ATP) production, leading to the activation of the adenosine monophosphate (AMP) -activated protein kinase pathway and subsequent inhibition of mTOR pathway (Head et al., 2015).

Testing Itraconazole on experimental settings was associated also with tumor hypoxia, as proved by induction of tumor-specific expression of Hypoxia-inducible factor 1-alpha (HIF1α), as well as decreased tumor micro-vessel load.

Taken together, these data support that Itraconazole may become a promising novel anti-angiogenic agent and In contrast to bevacizumab, Itraconazole is an inexpensive oral agent, currently available in a generic formulation and has been safely administered to thousands of patients as an antifungal drug with an excellent tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV NSCLC patients who have not received chemotherapy for metastatic disease management yet or inoperable locally recurrent Stage III NSCLC after concurrent chemoradiotherapy.
2. ECOG 0-2.
3. Age >18 years.
4. Adequate bone marrow reserve (white blood cells [WBC] ≥ 3.5 × 109 /L, neutrophils ≥ 1.5 × 109 /L, platelets ≥ 100 × 109 /L, and hemoglobin ≥ 9.0 gm/dL).

Exclusion Criteria:

1. Inadequate liver function (bilirubin > 1.5 times upper normal limit [ULN] and alanine transaminase [ALT] or aspartate transaminase [AST] > 3.0 ULN or up to 5.0 UNL in the presence of hepatic metastases).
2. Inadequate renal function (creatinine > 1.25 times ULN, creatinine clearance < 50mL/min).
3. Serious comorbid systemic disorder incompatible with the study.
4. Presence of other primary malignancy.
5. Patients with evidence of ventricular dysfunction such as congestive heart failure (CHF) or a history of CHF.
6. Patients with hypersensitivity to Itraconazole.
7. Patients receiving any Cytochrome P450 (CYP 3A4) inhibitor as clarithromycin, diltiazem, verapamil, quinidine ….etc.
8. Pregnant female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-12-02 (Estimated); Study Completion 2020-12-02 (Estimated)

PRIMARY OUTCOMES:
one year progression free survival | 1 year
  time from treatment initiation to either progression, death from any cause or lost to follow up.

SECONDARY OUTCOMES:
one year overall survival | 1 year
  time in months from time of diagnosis to death or date of last contact.
Radiological response | 18 weeks
  To compare radiological response of patients with advanced lung cancer receiving platinum bases chemotherapy combined with itraconazole to those receiving platinum based chemotherapy only after 3 and 6 cycles of chemotherapy.
quality of life | 18 weeks
  Patient's quality of life will be assessed at baseline, after 3 cycles, and at the end of chemotherapy treatment using EORTC modules specific to lung cancer.
Adverse effects of Itraconazole. | 18 weeks
  Incidence and severity will be evaluated using National Cancer Institute-Common Toxicity Criteria for adverse events (CTCAE V4.03).

CONTACTS AND LOCATIONS:
Overall Officials: Amr Shafik Tawfik, MD, Principal Investigator — oncology department at Ain shams University
Locations (1):
- oncology department Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
According to the sharing protocol of the official affliation

REFERENCES:
- [Derived] Mohamed AW, Elbassiouny M, Elkhodary DA, Shawki MA, Saad AS. The effect of itraconazole on the clinical outcomes of patients with advanced non-small cell lung cancer receiving platinum-based chemotherapy: a randomized controlled study. Med Oncol. 2021 Feb 9;38(3):23. doi: 10.1007/s12032-021-01475-0. PMID 33559053